CLINICAL TRIAL: NCT06930729
Title: Optimizing Care for Cancer Survivors With Depression (OASIS): Project 3
Brief Title: Optimizing Care for Cancer Survivors With Depression: Project 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Dahne, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00142262; R01CA281740 (NIH)
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Depression
MeSH Terms: conditions — Neoplasms; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digitally-Enhanced Stepped Care (Experimental): Participants randomized to the Digitally-Enhanced Stepped Care condition will be instructed to utilize a Behavioral Activation therapy focused mobile application called "Moodivate" regularly, at least once per day, for the treatment of depressed mood among cancer survivors. Participants in the Digitally-Enhanced Stepped Care group will receive a download code to download the Moodivate mobile application. Moodivate is a mobile app for individuals with elevated symptoms of depression. Within the app, users identify values, create activities, schedule activities, and rate mood daily. Participants will be asked to complete questionnaire measures at weeks 12, 16, 20, and 24 post-randomization. App engagement will be passively monitored for two weeks following initial download to determine whether care needs to be stepped up to guideline-concordant standard care.
  Interventions: Behavioral: Behavioral Activation Therapy App
- Guideline-Concordant Standard Care (Active Comparator): Participants randomized to the Guideline-Concordant Standard Care condition will receive 8 sessions of telehealth-delivered Behavioral Activation therapy with a mental health provider over a 10 week period. Participants will be asked to complete questionnaire measures at weeks 12, 16, 20, and 24 post-randomization.
  Interventions: Behavioral: Telehealth Delivered Behavioral Activation

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy App — Moodivate focuses on tracking daily activities, recording daily mood, and identifying new activities to complete that may help improve mood. Participants will be asked to complete questionnaire measures at weeks 12, 16, 20, and 24 post-randomization.
  Arms: Digitally-Enhanced Stepped Care
Behavioral: Telehealth Delivered Behavioral Activation — 8 sessions of telehealth-delivered Behavioral Activation with a mental health provider over a 10-week period.
  Arms: Guideline-Concordant Standard Care

SUMMARY:
The purpose of this research study is to evaluate different depression treatment approaches among cancer survivors. A cancer survivor is defined as anyone who is living and has been diagnosed with cancer.

Participants will be randomly assigned to either receive a mobile app for depression treatment, called "Moodivate", or to receive telehealth depression treatment sessions. Approximately 2/3 of participants enrolled will receive the mobile app and the remaining 1/3 will receive depression treatment via telehealth. Participants that receive Moodivate may later be assigned to also receive depression treatment via telehealth based their response to the Moodivate app. Participants will be asked to either use the Moodivate app and/or receive depression treatment via telehealth for a period of 10 weeks.

All participants will be asked to electronic questionnaire measures throughout the study period. Questionnaires will assess symptoms of depression, as well as general experiences using Moodivate and participating in this trial. Participation in this study will take about 24 weeks.

Participation in this study may help improve options for emotional wellness for cancer survivors. The greatest risks of this study include frustration, worsening of emotional distress, data breach, and/or loss of confidentiality.

DETAILED DESCRIPTION:
Depression is Highly Prevalent Among Cancer Survivors and Novel Care Delivery Approaches are Needed. Nearly one in four cancer survivors suffer from depression, with negative sequalae including lower quality of life, reduced adherence to cancer treatments, suicidal ideation, and desire for hastened death. Guidelines from leading oncology and mental health organizations including the American Society of Clinical Oncology (ASCO), the National Comprehensive Cancer Network, and the Commission on Cancer, recommend empirically based psychosocial interventions, such as Behavioral Activation (BA), as first line therapies. Unfortunately, despite guidelines, multilevel barriers, including transportation issues, stigma, and a scarcity of oncology mental health providers, limit widespread access to psychosocial first line depression therapies via usual care delivery approaches. These barriers are highly prominent in South Carolina (SC), the state at the focus of this Team Science Award. All SC counties contain medically underserved areas, and 15% of South Carolinians reside in rural areas. Novel care delivery approaches that address these multilevel barriers and extend psychosocial treatment access for cancer survivors in SC and beyond are clearly needed.

Self-guided digital mental health interventions (DMHIs) are an alternative psychosocial treatment delivery approach uniquely suited to addressing multilevel treatment barriers. Such interventions are delivered via technology-based platforms such as mobile apps, offer adaptations of evidence-based interventions, decrease the need for trained providers, and have a large evidence base in the general population as well as among cancer survivors indicating feasibility, acceptability, and comparable effects to standard psychosocial interventions when used as directed. Self-guided DMHIs are particularly well suited to the needs of cancer survivors because their flexible, self-directed pace can accommodate fluctuations in physical and mental health symptoms experienced due to cancer progression, side-effects, and/or cancer treatment transitions.

The extant literature on digital stepped care approaches has been similarly limited in terms of when and how decisions to step up care are made. Despite mounting evidence highlighting between-patient variability in DMHI engagement and clear, logical connection between engagement and clinical response, extant digitally-enhanced stepped care approaches have relied on clinical symptom change as the deciding factor for stepping. Whereas symptom change must be assessed over the course of months, intervention engagement can be assessed soon after starting treatment. By using passively collected DMHI analytics data, patients who do not engage with the DMHI can be stepped up, reducing delays in receipt of appropriate treatment. Evaluation of a stepped-care model, whereby cancer survivors with depressive symptoms first receive a low resource-intensive, yet still evidence-based, self-guided DMHI and then, if they do not engage within the first two weeks, are stepped up to the more resource-intensive gold standard psychosocial intervention, could help realize precision population health goals of providing the most effective and least resource-intensive intervention to all patients.

The current study will evaluate a digitally-enhanced stepped depression treatment approach for cancer survivors. This trial will lay the groundwork for a P01 project that will determine whether a digitally-enhanced stepped depression treatment approach for cancer survivors is non-inferior to guideline-concordant standard care in terms of depression treatment efficacy but superior for other key implementation outcomes (reach, cost-effectiveness, etc.). Our primary endpoint herein is feasibility of the stepped care approach among cancer survivors with elevated depressive symptoms. Secondarily, we will describe efficacy of the stepped care approach vs. guideline-concordant standard care.

ELIGIBILITY:
Inclusion Criteria:

* age 18+
* cancer survivor
* current elevated depressive symptoms defined per ASCO as a PHQ-9 score ≥ 8
* not currently receiving psychosocial depression treatment
* have the ability to complete treatment via telehealth and use Moodivate
* have a valid e-mail address or text message access (for assessments)
* English fluency

Exclusion Criteria:

- Current suicidal ideation at final eligibility screening (PHQ-9 item 9 ≥1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a digitally-enhanced stepped care approach to depression treatment among cancer survivors. | 24 weeks
  Feasibility will be defined as either use of the digital mental health intervention (DMHI) at least once per week for >4 weeks (for DMHI engagers) or attendance at >4 therapy sessions (for DMHI non-engagers). Digitally-enhanced stepped care will be considered feasible if >80% of participants meet feasibility benchmarks.

SECONDARY OUTCOMES:
Efficacy of digitally-enhanced stepped depression care as compared to guideline-concordant standard care among cancer survivors | 24 Weeks
  Descriptive change in Patient Health Questionnaire (PHQ-9) from baseline through 24 weeks in depressive symptoms as a function of randomization group.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dahne, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States